CLINICAL TRIAL: NCT01721447
Title: The Use of Optison Echocardiography Contrast in the Detection of Left Atrial Appendage Thrombus With Transesophageal Echocardiography.
Brief Title: Efficacy of Optison Echo Contrast to Detect Thrombus in Left Atrial Appendage
Acronym: DOLOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brent Wilson, Assistant Professor of Internal Medicine, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-OPT-018 GE
Record Dates: First submitted 2012-10-25; First posted 2012-11-05 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; stroke; TEE; Left atrial thrombus
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Echo arm (Experimental): Subjects with atrial fibrillation who are undergoing a TEE procedure will be assessed using Optison echocardiography contrast agent
  Interventions: Drug: Optison echocardiography contrast agent

INTERVENTIONS:
Drug: Optison echocardiography contrast agent — Subjects undergoing transesophageal echocardiography who will receive the Optison contrast agent during the procedure to test if the image quality improves to provide accurate assessment of the presence of left atrial thrombus.
  Other Names: Perflutren Protein-Type A microspheres

SUMMARY:
The investigators intend to determine if using Optison echocardiography contrast increases sensitivity and specificity of detecting left atrial appendage thrombus in transesophageal echocardiography studies as opposed to standard 2D and 3D TEE imaging without the use of echo contrast.

DETAILED DESCRIPTION:
Accurate determination of the presence or absence of left atrial appendage (LAA) thrombus has a large impact on the clinical course of patients with atrial fibrillation or ischemic stroke and has large financial implications as well. Misdiagnosing the presence of LAA thrombus can lead to unnecessarily cancelled procedures (cardioversion and atrial fibrillation ablation) and potentially hazardous, unnecessary changes in clinical care (such as prolonged Coumadin anticoagulation). Missing LAA thrombus can result in continuation of cardioversion or atrial fibrillation ablation procedures at a time when there is higher risk of subsequent embolic stroke.

Several of the patients with atrial fibrillation require transesophageal echocardiography (TEE) performed prior to cardioversion or atrial fibrillation ablation procedures. There is opportunity to enroll most of these patients in our proposed study. There has been essentially no work published about the use of echo contrast materials in TEE (other than agitated saline), particularly the use of Optison. Thus, the investigators will be exploring a new field in echocardiography and echo contrast.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Cognitively sound and able to provide informed consent
* Indicated for TEE as a standard clinical procedure for evaluation of cardiac health status.

Exclusion Criteria:

* Contraindicated for Optison administration
* Known right-to-left or bi-directional cardiac shunts
* Hypersensitivity to perflutren, blood, blood products or albumen
* Women who are pregnant
* Removal of Left Atrial Appendage
* Not able to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent D Wilson, MD, PHD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Wei K, Mulvagh SL, Carson L, Davidoff R, Gabriel R, Grimm RA, Wilson S, Fane L, Herzog CA, Zoghbi WA, Taylor R, Farrar M, Chaudhry FA, Porter TR, Irani W, Lang RM. The safety of deFinity and Optison for ultrasound image enhancement: a retrospective analysis of 78,383 administered contrast doses. J Am Soc Echocardiogr. 2008 Nov;21(11):1202-6. doi: 10.1016/j.echo.2008.07.019. Epub 2008 Oct 10. PMID 18848430
- [Background] Clark LN, Dittrich HC. Cardiac imaging using Optison. Am J Cardiol. 2000 Aug 17;86(4A):14G-18G. doi: 10.1016/s0002-9149(00)00984-x. PMID 10997346
- [Background] Bhatia VK, Senior R. Contrast echocardiography: evidence for clinical use. J Am Soc Echocardiogr. 2008 May;21(5):409-16. doi: 10.1016/j.echo.2008.01.018. Epub 2008 Mar 10. PMID 18329848
- [Background] Bednarz JE, Spencer KT, Weinert L, Sugeng L, Mor-Avi V, Lang RM. Identification of cardiac masses and abnormal blood flow patterns with harmonic power Doppler contrast echocardiography. J Am Soc Echocardiogr. 1999 Oct;12(10):871-5. doi: 10.1016/s0894-7317(99)70195-1. PMID 10511659

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Echo Arm
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Echo Arm
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 95
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Confidence in Assessment of Left Atrial Appendage Thrombus
Description: Confidence among echo readers to determine presence or absence of left atrial appendage thrombus before and after injection of Optison contrast agent. Percent confidence was calculated from a subjective assessment made by each reader after viewing the echo images. A six-point scale was used by the readers to grade the subjective assessment of their confidence in detecting thrombus; a score of 0 representing 0% (no confidence) up to a score of 5 representing 100% (total confidence) that the interpretation was correct for presence or absence of left atrial appendage thrombus. The reported percent confidence is the average of both echo readers.
Time Frame: One Transesophageal Echocardiography, up to 1 hour
Measure: Mean (Standard Deviation); unit: Percentage of Confidence
Groups:
- Pre-Contrast: Standard trans-esophageal echocardiography imaging prior to injection of Optison contrast
- Post-Contrast: Trans-esophageal echocardiography imaging following injection of Optison contrast
Arm/Group | Pre-Contrast | Post-Contrast
Number analyzed (Participants) | 100 | 100
Percentage of Confidence | 55 (12.5) | 95 (7.5)
Statistical Analysis 1: Comparison: Pre-Contrast vs Post-Contrast; Test type: Superiority; p < 0.001, Chi-squared

2. Secondary Outcome: Concordance Between Echo Readers in Determining Presence or Absence of Thrombus in the Left Atrial Appendage
Description: Percent agreement between echo readers to determine presence or absence of left atrial appendage thrombus before and after injection of Optison contrast agent
Time Frame: One transesophageal echocardiography, up to 1 hour
Measure: Number; unit: Percentage of Agreement
Arm/Group | Pre-Contrast | Post-Contrast
Number analyzed (Participants) | 100 | 100
Percentage of Agreement | 72 | 96
Statistical Analysis 1: Comparison: Pre-Contrast vs Post-Contrast; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Echo Arm
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Echo Arm (N=100)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT01721447/Prot_SAP_000.pdf